CLINICAL TRIAL: NCT07331285
Title: Bi-lateral HGN Therapy in Real-World Patients -Post Approval Research Investigation
Acronym: BREATHE
Status: Not yet recruiting | Type: Observational
Sponsor: Nyxoah Inc. (Industry)
Responsible Party: Sponsor
Organization: Nyxoah S.A. (Industry)
Other Study IDs: CL-BREATHE-2025
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; Hypoglossal Nerve Stimulation; Genio; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Genio System 2.1: This is a single-arm study. All consented and eligible subjects will be implanted with the Genio 2.1 System.
  Interventions: Device: This is a single arm study, all consented and eligible subjects will be implanted with the Genio® System 2.1

INTERVENTIONS:
Device: This is a single arm study, all consented and eligible subjects will be implanted with the Genio® System 2.1 — Genio® System 2.1
  Other Names: Genio Therapy

SUMMARY:
The objective of the BREATHE study is to demonstrate the continued safety and effectiveness of the Genio® System in treating subjects diagnosed with moderate to severe obstructive sleep apnea (OSA) who are intolerant to or failed/refused PAP treatments.

DETAILED DESCRIPTION:
BREATHE is a multicenter, prospective, single-arm, post-approval study. Following a baseline visit and implantation of the Genio® System 2.1, subjects will be asked to return for a therapy activation visit at approximately 8 weeks post-implant surgery.

The subject will have follow-up visits at 6 months, 9 months, 12 months and every 6-months thereafter up to 5 years post-implant surgery. Additional visits (for device titration or other reasons) are per standard of care and at the Investigator's discretion. Endpoints will be assessed at 12, 24, 36, 48 and 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Have an apnea-hypopnea index (AHI) greater than or equal to 15 and less than or equal to 65, measured on a full-night PSG performed no earlier than 2 years prior to enrollment (AHI4 and ODI4 available).
2. Be adults 22 years of age and older.
3. Have been confirmed to have failed, not tolerated, or be ineligible to be treated with current standard of care treatments for moderate to severe OSA.
4. Have pursued insurance pre-authorization for Genio® Therapy, recognizing that pre-authorization does not ensure payment, or demonstrate willingness to assume any out-of-pocket costs. The sponsor will not be responsible for treatment-related charges.
5. Agree to participate in the study and voluntarily sign and date an informed consent form.
6. Be willing and capable of complying with all study requirements, including specific lifestyle considerations, performing all follow-up visits, evaluation procedures and questionnaires for the whole duration of the trial.
7. Have a result of a Drug- Induced Sleep Endoscopy (DISE), no earlier than 2 years prior to enrollment.

Exclusion Criteria:

1. Combined central and mixed apnea-hypopnea index (AHI) greater than or equal to 25% of the total AHI.
2. Any functional or structural problem, medical illness or condition that would prevent or interfere with implantation, activation or continued use of the Genio® Therapy.
3. Have an implantable device which may be susceptible to unintended interaction with the Genio® System 2.1.
4. Women who are pregnant, planning to become pregnant or breastfeeding.
5. Any condition or procedure that has compromised neurological control of the upper airway.
6. Be part of the populations for which the safety and effectiveness of the Genio® System 2.1 has not been fully assessed:

   1. Patients below 22 or above 75 years of age.
   2. Patients with a Body Mass Index (BMI) above 32 kg/m2.
   3. Patients with an Apnea Hypopnea Index (AHI) below 15 or over 65 events/hr.
   4. Patients with Complete Concentric Collapse (CCC) at the soft palate level.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with moderate to severe obstructive sleep apnea (OSA) who are intolerant to or failed/refused PAP treatments.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Change in Apnea Hypopnea Index (AHI4%) | 12 months
  Percentage of responders at 12 months based on AHI4
Change in Oxyhemoglobin Desaturation Index (ODI4%) | 12 months
  Percentage of responders at 12 months based on ODI4
Device related SAEs | 12 months
  Incidence of device-related Serious Adverse Events at 12 months post-surgery
Device-related and procedure-related SAEs | 12 months
  Incidence of device-related and procedure-related SAEs at 12 months post-surgery

SECONDARY OUTCOMES:
Mean change in AHI4 | Baseline to 5 years
  Mean change in AHI4 from screening to 12, 24, 36, 48, and 60 months post-surgery.
Mean change in ODI4 | Baseline to 5 years
  Mean change in ODI4 from screening to 12, 24, 36, 48, and 60 months post-surgery.
% responders AHI4 | 2 years through 5 years
  Percentage of responders at 24, 36, 48, and 60 months based on AHI4 according to "Sher criteria".
% responders ODI4 | 2 years through 5 years
  Percentage of responders at 24, 36, 48 and 60 months based on ODI4
Subject Satisfaction | 1 year through 5 years
  Subject reported satisfaction with therapy (measured via bespoke questionnaire) measured at 12, 24, 36, 48, and 60 months post-surgery
Improvement in ESS | 1 year through 5 years
  Improvement in OSA-related symptoms (measured via Epworth Sleepiness Scale (ESS) questionnaire) measured at 12, 24, 36, 48, and 60 months post-surgery
Change in health status | 1 year through 5 years
  Subject reported impression of change in health status (measured via Patient Global Impression of Change (PGIC) questionnaire) at 12, 24, 36, 48, and 60 months post-surgery.
Clinician impression of change in Subject's health status | 1 year through 5 years
  Clinician impression of change in Subject's health status (measured via Clinician Global Impression of Change (CGIC) questionnaire) at 12, 24, 36, 48, and 60 months post-surgery.
Device-related Serious Adverse Events | 2 years through 5 years
  Incidence of device-related Serious Adverse Events, as reported by Investigator and adjudicated by the CEC, at 24, 36, 48, and 60 months post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Nyxoah, Inc, Summit, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woodson BT, Kent DT, Huntley C, Hancock MK, Van Daele DJ, Boon MS, Huntley TC, Mickelson S, Gillespie MB, Suurna MV, Kacker A, Roy A, MacKay S, Withrow KP, Dedhia RC, Huyett P, Heiser C, Nicola SD, Makori F, Vanderveken OM, Padyha TA, Magalang UJ, Chio E, Kezirian EJ, Lewis R. Bilateral hypoglossal nerve stimulation for obstructive sleep apnea: a nonrandomized clinical trial. J Clin Sleep Med. 2025 Nov 1;21(11):1883-1891. doi: 10.5664/jcsm.11822. PMID 40702817